CLINICAL TRIAL: NCT02035956
Title: First-in-human Study Evaluating the Safety, Tolerability and Immunogenicity of i.n. Administration of a Personalized Vaccination With IVAC MUTANOME Vaccine w/o Initial Treatment With RBL001/RBL002 Vaccine in Patients With Advanced Melanoma
Brief Title: IVAC MUTANOME Phase I Clinical Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech RNA Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Organization: BioNTech SE (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB_0004-01
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Melanoma
Keywords: IVAC MUTANOME; IVAC; personalized therapy; personalized immuno therapy; RB_0004-01; Ribological; Melanoma; cancer vaccine
MeSH Terms: conditions — Melanoma | interventions — Cancer Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IVAC MUTANOME RBL001/RBL002 (Experimental): All participants will be treated with the personalized IVAC MUTANOME vaccine with or without prior treatment with RBL001/RBL002 vaccine depending on expression of these two antigens. Vaccines will be administered intra-nodally.
  Interventions: Biological: IVAC MUTANOME, RBL001/RBL002

INTERVENTIONS:
Biological: IVAC MUTANOME, RBL001/RBL002 — Each patient will receive multiple repeated intranodal injections of IVAC MUTANOME vaccine with or without initial treatment with RBL001/RBL002.
  Other Names: cancer vaccine

SUMMARY:
Clinical first-in-human study evaluating the safety, tolerability and immunogenicity of intra-nodal administration of a personalized vaccination with IVAC MUTANOME vaccine with or without initial treatment with RBL001/RBL002 vaccine in patients with advanced melanoma

DETAILED DESCRIPTION:
IVAC MUTANOME is a poly-neo-epitopic coding RNA vaccine targeting the unique mutation signature of an individual patient. It is engineered on demand, provided as two patient-specific RNA drug products and administered as an individual treatment.

RBL001/RBL002 and IVAC MUTANOME are naked ribonucleic acid (RNA) based recombinant vaccines optimized to induce antigen-specific CD8+ and CD4+ T cell responses against melanoma associated target antigens.

The two antigens are well characterized antigens in melanoma that have been previously utilized with excellent safety and proven immunogenicity as vaccine targets in a number of independent clinical trials.

The overall rationale of the study is to determine safety of the novel RNA-based vaccine strategy and determine the number and function of vaccine-induced antigen-specific immune-responses as early biomarkers for the clinical mode of action.

The IVAC MUTANOME vaccine approach is based on targeting multiple immunogenic tumour mutations unique to a given patient's tumour using a poly-epitopic RNA-based vaccine manufactured for use in a single patient only. Parallel to the target discovery process and on demand manufacturing of IVAC MUTANOME vaccine patients with RBL001 and/ or RBL002 positive-tumours will receive the RBL001/RBL002 vaccine. Patients which tumours that are RBL001 and RBL002 negative can also be included into the clinical study but will not receive RBL001/RBL002 prior to IVAC MUTANOME. Applying this approach the RBL001/RBL002 vaccine and the IVAC MUTANOME vaccine administration is expected to lead to several effects contributing to their immunological (therapeutic) effects.

ELIGIBILITY:
Inclusion Criteria:

* Malignant Melanoma, resectable stage IIIA-C and IV (AJCC 2009 melanoma classification)
* Patients with unresectable Malignant Melanoma stage IIIA-C in complete remission, partial remission or stable disease after treatment with vemurafenib or patients with slow progressive disease.
* Malignant Melanoma, unresectable stage IV (AJCC 2009 melanoma classification) in complete remission, partial remission or stable disease after treatment with vemurafenib
* All lines of treatment for malignant melanoma are accepted.
* First line therapy for subjects not eligible or declining other first line therapies after all available treatment options have been transparently disclosed (to be documented in patient medical record).
* ≥ 18 years of age
* Written informed consent
* ECOG performance status (PS) 0-1 (appendix G)
* Life expectancy > 6 months
* WBC ≥ 3x109/L
* Haemoglobin ≥ 10 g/dl
* Platelet count ≥ 100,000/mm³
* LDH level < 2.0 x ULN
* Negative pregnancy test (measured by β-HCG) for females which are childbearing potential
* Suitable lymph nodes for injection using ultrasound guidance

Exclusion Criteria:

* Pregnancy or breastfeeding
* Primary ocular melanoma
* History (< 5 years) of a second malignancy other than squamous or basal cell carcinoma, non-active prostate cancer or cervical carcinoma in situ
* Brain metastases
* Known or symptomatic pleural effusions and/or ascites
* Known hypersensitivity to the active substance or to any of the excipients
* A serious local infection (e.g. cellulitis, abscess) or systemic infection (e.g. pneumonia, septicemia) which requires systemic antibiotic treatment within 2 weeks prior to the first dose of study medication
* Positive test for acute or chronic active hepatitis B or C infection, acute EBV or acute CMV injection
* Clinically relevant autoimmune disease
* Systemic immune suppression:
* HIV disease
* Use of chronic oral or systemic steroid medication (topical or inhalational steroids are permitted)
* Other clinical relevant systemic immune suppression
* Symptomatic congestive heart failure (NYHA 3 or 4)
* Unstable angina pectoris
* Radiotherapy within two weeks, myelosuppressive chemotherapy, ipilimumab and major surgery within 4 weeks/28 days before the first treatment. Interferon and approved BRAF inhibitors will be allowed as concurrent treatment.
* Any investigational drug within 4 weeks/28 days or 5 half-lives depending on what gives the longer range before the first treatment of this study
* Minor surgery within 14 days before the first treatment of this study
* Fertile males and females who are unwilling to use a highly effective method of birth control (less than 1% per year, e.g. condom with spermicide, diaphragm with spermicide, birth control pills, injections, patches or intrauterine device) during study treatment and 28 days after the last dose of study treatment
* Presence of a serious concurrent illness or other condition (e.g. psychological, family, sociological, or geographical circumstances) that does not permit adequate follow-up and compliance with the protocol

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of repetitive doses | up to a maximum of 189 days
  Number of Patients with adverse events, total number of adverse events

SECONDARY OUTCOMES:
Monitoring of vaccine-induced cellular immune response, | 161 days
  Determination of pharmacodynamic activity

CONTACTS AND LOCATIONS:
Overall Officials: Ugur Sahin, Prof. Dr., Study Director — BioNTech RNA Pharmaceuticals GmbH
Locations (3):
- Medizinische Universität Wien, Vienna, AT-Wien, Austria
- Germany (2):
  - Hautklinik und Poliklinik Universitätsmedizin der Johannes-Gutenberg Universität Mainz, Mainz
  - Klinik für Dermatologie, Venerologie und Allergologie UMM - Universitätsmedizin Mannheim Medizinische Fakultät Mannheim der Ruprecht-Karls-Universität Heidelberg, Mannheim

REFERENCES:
- [Derived] Weber D, Ibn-Salem J, Sorn P, Suchan M, Holtstrater C, Lahrmann U, Vogler I, Schmoldt K, Lang F, Schrors B, Lower M, Sahin U. Accurate detection of tumor-specific gene fusions reveals strongly immunogenic personal neo-antigens. Nat Biotechnol. 2022 Aug;40(8):1276-1284. doi: 10.1038/s41587-022-01247-9. Epub 2022 Apr 4. PMID 35379963